CLINICAL TRIAL: NCT05155189
Title: A Clinical Study to Evaluate Safety and Efficacy of C-CAR031 Armored CAR-T Cell Injection in Treatment of Advanced Hepatocellular Carcinoma
Brief Title: A Study to Evaluate Safety and Efficacy of Armored CAR-T Cell Injection C-CAR031 in Advanced Hepatocellular Carcinoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, TingBo Liang, professor, Zhejiang University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0921-028
Record Dates: First submitted 2021-12-07; First posted 2021-12-13 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Hepatocellular Carcinoma
Keywords: Liver Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — lenvatinib; regorafenib; durvalumab

STUDY DESIGN:
Intervention Model Description: Four Groups Assignment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- C-CAR031 (Experimental): Autologous C-CAR031 administered by intravenous (IV) infusion
  Interventions: Biological: C-CAR031
- C-CAR031 combined with Lenvatinb (Experimental): Autologous C-CAR031 combination with Lenvatinib
  Interventions: Biological: C-CAR031; Drug: Lenvatinib
- C-CAR031 combined with Regorafenib (Experimental): Autologous C-CAR031 combination with Regorafenib
  Interventions: Biological: C-CAR031; Drug: Regorafenib (BAY 73-4506)
- C-CAR031 combined with Durvalumab (Experimental): Autologous C-CAR031 combination with Durvalumab
  Interventions: Biological: C-CAR031; Drug: Durvalumab

INTERVENTIONS:
Biological: C-CAR031 — Targeting GPC3 armored CART cell injection (C-CAR031)
Drug: Lenvatinib — Tyrosine kinase inhibitors
  Arms: C-CAR031 combined with Lenvatinb
Drug: Regorafenib (BAY 73-4506) — Tyrosine kinase inhibitors
  Arms: C-CAR031 combined with Regorafenib
Drug: Durvalumab — Immune checkpoint inhibitors, ICIs
  Arms: C-CAR031 combined with Durvalumab

SUMMARY:
A study that aimed to assess the safety and anti-tumor activity of CCAR031 injection in unresectable HCC patients.

DETAILED DESCRIPTION:
This study plans to enroll 4-36 patients to assess the safety of C-CAR031. Subjects who meet the eligibility criteria will receive a single dose of C-CAR031 injection, and will be followed up post-treatment for safety monitoring. This study will also enroll 6-36 patients to further explore the treatment modality of combination with Lenvatinib, Regorafenib or Durvalumab at explored safe and effective dose level(s) of C-CAR031 monotherapy in specific eligible advanced HCC patients to provide data support for the phase II study of CAR-T combination therapy. The follow-up period will be 12 months.

ELIGIBILITY:
Inclusion Criteria:

* 1.Voluntary participation and able to sign the informed consent form
* 2. Aged 18 to 75 years at screening
* 3. Patients with histologically confirmed hepatocellular carcinoma (HCC) who meet the following requirements: a. Barcelona Clinic Liver Cancer Stage B or C (BCLC B/C) b. Child-Pugh score ≤ 6 c. GPC3 is possibly expressed in tumor tissues
* 4. Patients with relapsed / progressive disease after at least one prior standard systemic therapy for HCC, or ineligible to accept/unable to tolerate the systemic therapies. Standard systemic therapies may include targeted drugs (such as Sorafenib, Lenvatinib, Donafenib, Apatinib), immune checkpoint inhibitors (such as Atezolizumab, Pembrolizumab, Camrelizumab, Sintilimab, Nivolumab, Toripalimab, Tislelizumab) or chemotherapeutic drugs (such as Oxaliplatin and 5-Fu). Subjects in theC-CAR031 plus Lenvatinib group must meet the following criteria: (1)have not received prior Lenvatinib therapy; (2) Progression or intolerance to one prior line of systemic therapy containing both immune checkpoint inhibitors and VEGF/VEGFR- targeted agents. Subjects in the C-CAR031 combination with Regorafenib group must meet the following criteria: (1)have not received prior Regorafenib therapy; (2) Progression or intolerance to one prior line of systemic therapy containing both immune checkpoint inhibitors and VEGF/VEGFR- targeted agents. Subjects in theC-CAR031 plus Durvalumab group must meet the following criteria:(1) Progression or intolerance to one prior line of systemic therapy containing both immune checkpoint inhibitors and VEGF/VEGFR-targeted agents; (2) no prior immune-related toxicity leading to permanent discontinuation of immunotherapy;(3) no history of ≥ Grade 3 immune-related adverse events (irAEs), or any grade immune-related neurological/ocular AEs. (Note: Subjects with ≤ Grade 2 endocrine AEs may enroll if asymptomatic on stable replacement therapy, excluding those: a. requiring non-corticosteroid immunosuppressants, b. experiencing AE recurrence upon immunotherapy rechallenge, c. or using corticosteroids at >10 mg/day prednisone or equivalent.) (4) All AEs associated with prior immunotherapy must have resolved or returned to pre-treatment levels prior to screening; (5) Body weight more than 30 kg.
* 5. At least one measurable target lesion (as per RECIST v1.1)
* 6. WHO/ECOG performance status (PS) score of 0 or 1 point
* 7. Expected survival ≥ 12 weeks
* 8. Left ventricular ejection fraction (LVEF) by echocardiography ≥ 45%
* 9. No active pulmonary infection; no known history of pneumonitis requiring steroids; absence of acute onset or progressive pneumonitis at baseline.
* 10. Laboratory tests: a. Absolute neutrophil count (ANC) ≥ 1.0 × 109/L b. Lymphocyte count ≥ 0.4 × 109/L c. Platelet count ≥ 60 × 109/L d. Hemoglobin ≥ 80 g/L e. Total bilirubin (TBIL) ≤ 2 × upper limit of normal (ULN) f. AST and ALT ≤ 5 × ULN g. Serum creatinine ≤ 1.5 × ULN h. Prothrombin time (PT): prolonged PT ≤ 4 s
* 11. Patients without history of HBV infection, or with HBV DNA < 2000 IU/mL (or 10000 copies/mL) at screening who agree to receive anti-virus therapies throughout the study according to the guidelines
* 12. Negative serum or urine pregnancy test results for females of child-bearing age at screening; In addition, they should agree to take effective contraceptive measures throughout the study
* 13. Patients who agree to abstain from drinking throughout the study

Exclusion Criteria:

* 1. History of severe allergic or hypersensitivity to DMSO. Subjects with known allergies to the active components of Lenvatinib, Regorafenib, or Durvalumab will be excluded from respective combination treatment groups.
* 2. History of liver transplantation
* 3. History of prior cell therapy
* 4. Tumor volume > 50% of the liver.
* 5. portal stem vein tumor thrombus
* 6. Moderate to severe ascites.
* 7. Metastases to bones or central nervous system (CNS), or involved CNS diseasesincluding hepatic encephalopathy, epilepsy, cerebrovascular accidents, etc.
* 8. Receipt of radiotherapy within 6 weeks prior to apheresis
* 9. Receipt of Local therapy (such as surgery, ablation, and intervention) within 4 weeks prior to apheresis or presence of unhealed wounds before apheresis
* 10. Receipt of systemic treatment and failure to meet the minimum requirements for wash-out periods before apheresis: a. Immune checkpointinhibitors: 2 weeks; b. Small molecule target therapy: < 7 days; c. Systemic anti-tumor therapies using experimental anticancer drugs or other Chinese herbal medicines and Chinese patent medicines with unclear mechanisms: 2 weeks; d. Steroids (except inhaled steroids) or other immunomodulators (including interleukins, interferons, and thymosins) of systemic therapeutic dose: 2 weeks; e. Any unresolved toxicity ≥ NCI CTCAE Grade 2 from prior anticancer therapy, except alopecia, vitiligo, and laboratory abnormalities explicitly permitted by the inclusion criteria.
* 11. Other history of primary cancers, excluding:a. Nonmelanoma skin cancer cured by resection (such as basal cell carcinoma) b. Cured carcinoma in situ (such as cervical cancer, bladder cancer, and breast cancer)
* 12. Active hepatitis C virus infection (HCV RNA positive)
* 13. Syphilis infection
* 14. History of active/immunodeficient diseases (including but not limited to HIV, systemic lupus erythematosus, inflammatory bowel disease, rheumatoid arthritis, myasthenia gravis, Graves' disease, and hypophysitis; excluding: vitiligo or alopecia, hypothyroidism in patients with stable medical conditions after hormone replacement therapy, any chronic skin conditions that need no systemic treatment, and other diseases judged by the investigator to be of no clinical significance)
* 15. Persistent and active infections (excluding prophylactic anti-infectives)
* 16. Uncontrolled hypertension, diabetes, arrhythmia, and symptomatic congestive heart failure
* 17. Dementia or mental state changes supported by obvious clinical evidence
* 18. Cardiac insufficiency: class III or IV, according to the New York Heart Association (NYHA) functional classifications
* 19. Unstable heart or lung diseases
* 20. Obvious bleeding risks or tendencies
* 21. Females who are pregnant or breastfeeding or expect to be pregnant or breastfeeding during the study
* 22. Other diseases that may add further risks to the subject or interfere with the study results as judged by the investigators
* 23. For combination with Lenvatinib, Regorafenib or Durvalumab, the following will be excluded: a. History of renal disease or nephrotic syndrome; b. Refractory nausea and vomiting, chronic gastrointestinal disease, inability to swallow formulation, or previous intestinal resection that precludes adequate absorption, distribution, metabolism, or excretion of Lenvatinib or Regorafenib; c. History of ≥ Grade 3 bleeding disorder, vasculitis, or significant gastrointestinal bleeding episodes within 28 days prior to screening; d. History of arterial thromboembolic events (ATEs), including myocardial infarction, cerebrovascular accident, or transient ischemic attack within 6 months prior to screening; e. Serious or non-healing wound, active gastrointestinal ulcer, or bone fracture within 28 days prior to screening; f. Use of full-dose anticoagulants or thrombolytics for non-prophylactic purposes within 10 days prior to screening; g. History of deep vein thrombosis, pulmonary embolism, or any other clinically significant thromboembolism within 3 months prior to screening; h. Presence of symptomatic or uncontrolled hypertension.
* 24. Uncontrolled intermittent severe chronic gastrointestinal disorders associated with diarrhea (excluded from the durvalumab treatment group).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2022-02-21 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2041-05 (Estimated)

PRIMARY OUTCOMES:
TEAEs | start pretreatment to 12 months
  treatment emergent adverse events
AESIs | start pretreatment to 12 months
  adverse events of special interest

SECONDARY OUTCOMES:
objective response rate by RECIST 1.1 | at Weeks 6, 12, and 18 and Months 6, 9, and 12 after cell infusion
  objective response rate according to RECIST 1.1
disease control rate by RECIST 1.1 | at Weeks 6, 12, and 18 and Months 6, 9, and 12 after cell infusion
  disease control rate according to RECIST 1.1
duration of response by RECIST 1.1 | at Weeks 6, 12, and 18 and Months 6, 9, and 12 after cell infusion
  duration of response according to RECIST 1.1
progression-free survival by RECIST 1.1 | The efficacy is evaluated at Weeks 6, 12, and 18 and Months 6, 9, and 12 after cell infusion.-
  progression-free survival to RECIST 1.1
objective response rate by mRECIST | The efficacy is evaluated at Weeks 6, 12, and 18 and Months 6, 9, and 12 after cell infusion.-
  objective response rate according to mRECIST
disease control rate by RECIST | The efficacy is evaluated at Weeks 6, 12, and 18 and Months 6, 9, and 12 after cell infusion.-
  disease control rate according to mRECIST
duration of response by mRECIST | The efficacy is evaluated at Weeks 6, 12, and 18 and Months 6, 9, and 12 after cell infusion.-
  duration of response according to mRECIST
progression-free survival by mRECIST | The efficacy is evaluated at Weeks 6, 12, and 18 and Months 6, 9, and 12 after cell infusion.-
  progression-free survival to mRECIST
overall survival | start pretreatment to the date of deaths
  overall survival
6-months overall survival | start pretreatment to 6 months after cell infusion
  6-months overall survival
12-months overall survival | start pretreatment to 12 months after cell infusion
  12-months overall survival

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - the First Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - The first affiliated hospital of Zhengzhou University, Zhengzhou

IPD SHARING:
Plan to Share IPD: No